CLINICAL TRIAL: NCT01735864
Title: Evaluation of the Efficacy and Safety of Indigo Naturalis Extract in Oil in the Topical Therapy of Psoriasis Vulgaris: Dosage Determination
Brief Title: Dosage Determination Trial for Indigo Naturalis Extract in Oil Ointment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yin-ku Lin, MD., PhD., Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSC101-2325-B-182-018
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis Vulgaris
Keywords: Indigo naturalis extract in oil
MeSH Terms: interventions — indirubin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Indirubin 200 μg/g (Active Comparator): per gram of ointment contains 200 μg of indirubin
  Interventions: Drug: Indirubin 200μg/g
- Indirubin 100 μg/g (Active Comparator): per gram of ointment contains 100 μg of indirubin
  Interventions: Drug: Indirubin 100 μg/g
- Indirubin 50 μg/g (Active Comparator): per gram of ointment contains 50 μg of indirubin
  Interventions: Drug: Indirubin 50 μg/g
- Indirubin 10 μg/g (Active Comparator): per gram of ointment contains 10 μg of indirubin
  Interventions: Drug: Indirubin 10 μg/g

INTERVENTIONS:
Drug: Indirubin 200μg/g — 1. Dosage form: Ointment
  2. Dose(s): Each gram of ointment containing 200 μg of indirubin
  3. Dosing schedule: apply 0.5 g of ointment per 10 x 10 cm psoriatic lesion twice daily
  Other Names: INEO ointment: Indirubin 200 μg/g
  Arms: Indirubin 200 μg/g
Drug: Indirubin 100 μg/g — 1. Dosage form: Ointment
  2. Dose(s): Each gram of ointment contains 100 μg of indirubin
  3. Dosing schedule: apply 0.5 g of ointment per 10 x 10 cm psoriatic lesion twice daily
  Other Names: INEO ointment: Indirubin 100 μg/g
  Arms: Indirubin 100 μg/g
Drug: Indirubin 50 μg/g — 1. Dosage form: Ointment
  2. Dose(s): Each gram of ointment contains 50 μg of indirubin
  3. Dosing schedule: apply 0.5 g of ointment per 10 x 10 cm psoriatic lesion twice daily
  Other Names: INEO ointment: Indirubin 50 μg/g
  Arms: Indirubin 50 μg/g
Drug: Indirubin 10 μg/g — 1. Dosage form: Ointment
  2. Dose(s): Each gram of ointment contains 10 μg of indirubin
  3. Dosing schedule: apply 0.5 g of ointment per 10 x 10 cm psoriatic lesion twice daily
  Other Names: INEO ointment: Indirubin 10 μg/g
  Arms: Indirubin 10 μg/g

SUMMARY:
The use of refined indigo naturalis (indigo naturalis extract in oil, INEO)ointment to treat psoriasis has been proven effective in our previous study. This study aims to evaluate the efficacy and safety of INEO ointment, and further determine the optimal concentration of INEO ointment (per gram of ointment containing either 200 μg, 100 μg, 50 μg or 10 μg of indirubin) in treatment of various local skin signs and thickness of psoriasis plaque.

DETAILED DESCRIPTION:
The use of indigo naturalis ointment to treat psoriasis has been proven effective in our previous clinical studies which demonstrated the efficacy and safety of topical indigo naturalis ointment, showing its ability to provide significant improvement of psoriatic skin lesions.

We developed a new formulation in which indigo naturalis powder is refined and reduces the blue discoloration of skin and clothes, making the treatment more user-friendly. We had observed an equivalent efficacy of the refined form of indigo naturalis (INEO) ointment on treating psoriasis as the crude form. However, it is necessary to determine an appropriate dosage of the refined form regarding its efficacy and safety.

This is a double-blind, 4-arm parallel study. The aim of this study is

1. To determine an appropriate dosage of indirubin in INEO ointment, regarding its efficacy and safety.
2. To evaluate the efficacy of INEO ointment in different local skin signs of plaque lesions.
3. To evaluate the efficacy of INEO in different traditional Chinese medicine clinical syndromes of psoriasis vulgaris.
4. To investigate the effects of INEO ointment on the immune system.
5. To evaluate the effects of INEO ointment in improving quality of life after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 - 65 years, men or women.
* Diagnosed as mild to moderate plaque-type psoriasis by the dermatologist, with psoriasis for a minimum of 1 year.
* Plaque psoriasis involving <20% of BSA and with PASI <20.
* Female patients of child-bearing age with negative pregnancy test at screening.
* Female patients of childbearing age who have agreed to continue using birth control measures approved by the investigator and agree not to lactate for the duration of the study.
* Willingness to comply with study protocol.
* With signed informed consent form.

Exclusion Criteria:

* With history of topically or systematically hypersensitive to indigo naturalis or its excipient in ointment.
* With history of sensitivity to Chinese herb.
* Received systematic treatment for psoriasis within 4 weeks.
* Received topical treatment for psoriasis within 2 weeks.
* With abnormal liver or renal function, clinically significant abnormalities in hematology, severe uncontrolled metabolic syndrome,psychiatric disease, cancer or AIDS.
* Patients with pustular or erythrodermic psoriasis.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Compare the mean percentage change of Psoriasis Areas Severity Index (PASI) from baseline at week 8 between groups | 8 weeks
  1. Mean change of total score (range 0-72)
  2. Percentage change of PASI
  3. Individual scores of scaling, erythema, and elevation by sites
  4. Percentage of responder (>50% of improvement, defined as clinical meaningful) and non-responder (less then 50% of improvement)
  5. Percentage of subjects achieving "clear or almost clear" (defined as PASI >90% of improvement)

SECONDARY OUTCOMES:
Body surface area (BSA)involved | 8 weeks
  1. Compare the BSA involved change from baseline on target psoriatic lesion(cm2)
  2. Compare the percentage change from baseline on target psoriatic lesion
Psoriasis Severity Index (PSI) | 8 weeks
  1. Mean change of total score (range 0-12) of the target psoriatic plaque
  2. Percentage change of PSI score of the target psoriatic plaque
  3. Clearing percentage of target psoriatic plaque (the target plaque before treatment is defined as 100%, and the clearance of lesion is defined as 0%)
Efficacy in various local skin signs | 8 weeks
  1. Thickness: thin (<0.05 mm), intermediate (≥0.05 to <1.0 mm) or thick (≥1.0 mm)
  2. Size: small (<5 cm in diameter), large (>5 cm in diameter) or concurrent (i.e., two type sizes exist)
  3. Erythema (redness): light red (ruddier (light red) than peripheral normal skin) or dark red (redder (scarlet) than peripheral normal skin)
Efficacy in different traditional Chinese medicine (TCM) clinical syndromes of psoriasis by PASI/PSI: | 8 weeks
  1. Blood-heat (血熱) syndrome
  2. Blood-dryness (血燥) syndrome
  3. Blood-stasis (血瘀) syndrome
Physician's Global Assessment (PGA) | 8 weeks
  0 = no sign of psoriasis, 1 = almost clear, 2 = mild, 3 = moderate, 4 = moderate to severe, and 5 = severe
Subject's Global Assessment (SGA) | 8 weeks
  0 = cleared, 1 = excellent, 2 = good, 3 = fair, 4 = poor, and 5 = worse
Dermatology Life Quality Index (DLQI) questionnaire | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Ku Lin, MD., PhD., Principal Investigator — Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital at Keelung
Locations (3):
- Taiwan (3):
  - Chang Gung Memorial Hospital at Keelung, Keelung
  - Chang Gung Memorial Hospital at Taipei, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan